CLINICAL TRIAL: NCT04739371
Title: Food Intake and Intra-Nasal Insulin for African American Adults
Brief Title: Food Intake and Intra-Nasal Insulin for African American Adults (FIINAAL)
Acronym: FIINAAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Nutrition Obesity Research Center (Other)
Responsible Party: Principal Investigator, Owen Carmichael, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PBRC 2020-047
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Insulin
Keywords: Intranasal Insulin; Food Intake; APOE; Cognition; African American
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin, Regular, Human; Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin (Experimental): 40 participants will receive 40 IUs of intranasal insulin about 30 minutes before consuming an ad libitum lunch.
  Interventions: Drug: Insulin, Regular, Human
- Placebo (Placebo Comparator): 40 participants will receive 40 IUs of intranasal saline about 30 minutes before consuming an ad libitum lunch.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin, Regular, Human — The spray will last a few seconds and then the participant will be asked to sniff to aid the drug into the nose. The device (i.e. ViaNase) is an atomizer that uses its patented technology that turns the liquid into a fine mist of droplets to facilitate the drug along the nose to brain pathway. Each nostril will receive this administration 2 times for a total of 40 IUs or 0.4 mL of liquid.
  Other Names: Novolin R
  Arms: Insulin
Drug: Placebo — The spray will last a few seconds and then the participant will be asked to sniff to aid the saline into the nose. The device (i.e. ViaNase) is an atomizer that uses its patented technology that turns the liquid into a fine mist of droplets to facilitate the drug along the nose to brain pathway. Each nostril will receive this administration 2 times for a total of 40 IUs or 0.4 mL of liquid.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this research study is to investigate brain insulin's relationship with food intake in African Americans. Facilitating insulin's entrance into the brain through a nasal spray is currently being studied as a way to prevent or treat Alzheimer's disease. However, brain insulin may also have an impact on food intake. This study is designed to help researchers understand how different factors related to Alzheimer's disease (i.e. APOE genotype and cognitive functioning) influence brain insulin's relationship with food intake.

DETAILED DESCRIPTION:
The investigators will utilize a double-blind, placebo-controlled, randomized crossover design comparing a single acute dose of intranasal insulin to a single acute dose of a saline placebo.

The primary aim will consist of exploring the differences in ingestive behaviors constructs (i.e. hunger, satiety, and fullness) and ad libitum lunch caloric intake between acute administration of either a dose of intranasal insulin or saline placebo. The hypothesis is that acute intranasal insulin will result in the consumption of fewer calories, greater feelings of satiety and fullness, and less hunger compared to acute saline. A secondary aim of this investigation will be to analyzing differences in food intake by APOE genotype, adiposity, and AD family history.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* are aged 45 years to 65 years old
* are willing to provide written informed consent
* speak and read English

Exclusion Criteria:

* diagnosed with type 1 or 2 diabetes
* pregnant or attempting to become pregnant
* have a history of sensitivity to glutaraldehyde

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Change in caloric intake | 30 minutes post intranasal insulin administration
  Caloric intake will be quantified by measuring the amount of the ad libitum lunch that is consumed. Caloric intake will be compared between insulin and placebo conditions to determine if caloric intake has increased or decreased.
Change in ingestive behavior constructs | 30 minutes post intranasal insulin administration
  Ingestive behavior constructs (e.g. hunger, satiety, fullness, etc.) will be quantified through the use of visual analogue scales that have a positive and negative rating at each end attached to a specific question to address each construct separately. Ingestive behavior outcomes will be compared between insulin and placebo conditions to determine if there are greater or lesser feelings of ingestive behavior constructs.

SECONDARY OUTCOMES:
Number of participants who are APOE e4 carriers versus noncarriers | Through study completion, an average of 1 year
  APOE genotype (i.e. APOE e4 carriers versus noncarriers) will be identified via blood assay.
Characterize AD family history (via a questionnaire) | Day 1
  AD family history, via a questionnaire, will be quantified by asking participants to identify immediate biological family members that have suffered from AD or dementia.
Amount of adiposity (i.e. DXA) per participant | Day 4
  Adiposity will be quantified via a DXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Owen T Carmichael, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data will be available upon request with the appropriate data transfer agreements established.
Time Frame: The data will be available after the primary results of the study have been published.
Access Criteria: By request